CLINICAL TRIAL: NCT04260438
Title: An Open-label, Randomized, Fed, Single Dose, Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerability of CKD-393 in Healthy Subjects
Brief Title: Clinical Study to Evaluate the Pharmacokinetics, Safety and Tolerability of CKD-393 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A98_01BE1922P
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lobeglitazone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): 1. Period 1: Treatment A
  2. Period 2: Treatment B
  3. Period 3: Treatment C
  Interventions: Drug: CKD-501 0.5mg Tab. 1T, D759 100mg Tab. 1T and D150 1000mg Tab. 1T; Drug: CKD-393 0.5/100/1000mg formulation 1 Tab. 1T; Drug: CKD-393 0.5/100/1000mg formulation 2 Tab. 1T
- Group 2 (Experimental): 1. Period 1: Treatment A
  2. Period 2: Treatment C
  3. Period 3: Treatment B
  Interventions: Drug: CKD-501 0.5mg Tab. 1T, D759 100mg Tab. 1T and D150 1000mg Tab. 1T; Drug: CKD-393 0.5/100/1000mg formulation 1 Tab. 1T; Drug: CKD-393 0.5/100/1000mg formulation 2 Tab. 1T
- Group 3 (Experimental): 1. Period 1: Treatment B
  2. Period 2: Treatment A
  3. Period 3: Treatment C
  Interventions: Drug: CKD-501 0.5mg Tab. 1T, D759 100mg Tab. 1T and D150 1000mg Tab. 1T; Drug: CKD-393 0.5/100/1000mg formulation 1 Tab. 1T; Drug: CKD-393 0.5/100/1000mg formulation 2 Tab. 1T
- Group 4 (Experimental): 1. Period 1: Treatment B
  2. Period 2: Treatment C
  3. Period 3: Treatment A
  Interventions: Drug: CKD-501 0.5mg Tab. 1T, D759 100mg Tab. 1T and D150 1000mg Tab. 1T; Drug: CKD-393 0.5/100/1000mg formulation 1 Tab. 1T; Drug: CKD-393 0.5/100/1000mg formulation 2 Tab. 1T
- Group 5 (Experimental): 1. Period 1: Treatment C
  2. Period 2: Treatment A
  3. Period 3: Treatment B
  Interventions: Drug: CKD-501 0.5mg Tab. 1T, D759 100mg Tab. 1T and D150 1000mg Tab. 1T; Drug: CKD-393 0.5/100/1000mg formulation 1 Tab. 1T; Drug: CKD-393 0.5/100/1000mg formulation 2 Tab. 1T
- Group 6 (Experimental): 1. Period 1: Treatment C
  2. Period 2: Treatment B
  3. Period 3: Treatment A
  Interventions: Drug: CKD-501 0.5mg Tab. 1T, D759 100mg Tab. 1T and D150 1000mg Tab. 1T; Drug: CKD-393 0.5/100/1000mg formulation 1 Tab. 1T; Drug: CKD-393 0.5/100/1000mg formulation 2 Tab. 1T

INTERVENTIONS:
Drug: CKD-501 0.5mg Tab. 1T, D759 100mg Tab. 1T and D150 1000mg Tab. 1T — single oral administration under fed condition
  Other Names: Treatment A
Drug: CKD-393 0.5/100/1000mg formulation 1 Tab. 1T — single oral administration under fed condition
  Other Names: Treatment B
Drug: CKD-393 0.5/100/1000mg formulation 2 Tab. 1T — single oral administration under fed condition
  Other Names: Treatment C

SUMMARY:
This study is an open-label, randomized, fed, single dose, crossover study to evaluate the pharmacokinetics, safety and tolerability of CKD-393 in healthy subjects

DETAILED DESCRIPTION:
To healthy subjects of twenty-four (24), following treatments are administered dosing in each period and wash-out period is a minimum of 7 days.

Reference drug: 1) CKD-501 0.5mg 2) D759 3) D150 Test drug: 1) CKD-393 0.5/100/1000mg formulation Ⅰ Tab. 2) CKD-393 0.5/100/1000mg formulation Ⅱ Tab.

Pharmacokinetic blood samples are collected up to 48hrs. The pharmacokinetic characteristics and safety are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, aged between ≥ 19 and ≤ 55 years old at the time of screening.
2. Weight ≥ 50kg, with calculated body mass index (BMI) of ≥ 18.5 and ≤ 29.9 kg/m2

   * BMI = Weight(kg)/ Height(m)2
3. Subject who consents to use at least two clinically effective birth controls for at least 1 month following the last dose.
4. Subject is informed of the investigational nature of this study and voluntarily agrees to participate in this study and comply with the relevant instructions in written.

Exclusion Criteria:

1. History or presence of clinically significant and sever active cardiovascular, respiratory, hepatobiliary, renal, endocrine, hematological, gastrointestinal, neurologic, immune, dermatologic or psychiatric disorder.
2. With symptoms indicating acute illness within 28 days prior to the first Investigational Product (IP) administration.
3. Any medical history that may affect drug absorption, distribution, metabolism and excretion.
4. Individuals who had history of hypersensitivity to follow drugs, derivative drugs or others drugs(aspirin and antibiotics etc.) or had history of drug abuse

   * Thiazolidinedione
   * DPP-4 inhibitor
   * Metformin
5. Any clinically significant chronic medical illness.
6. Any genetic disease including galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
7. Individuals with one of the following laboratory test results in screening

   * AST, ALT > UNL (upper normal limit) x 3
   * fasting glucose < 70 mg/dL or > 125 mg/dL
   * Creatinine clearance ≤ 80 mL/min
   * In ECG result, QTc > 450 msec
   * hCG(+) (only women)
8. Individuals who had positive test results at HBs Ag, anti-HCV Ab, anti-HIV Ab, VDRL.
9. Use of any prescription drugs within 14 days prior to study drug administration.
10. Use of over-the-counter medications and herbal preparations within 7 days prior to study drug administration.
11. History of any clinically significant allergic reaction (However, mild allergic rhinitis or allergic dermatitis which do not required medication may be allowed).
12. Individuals who cannot eat standard meal provided from clinical trial center.
13. Donation of blood within 60 days prior to study drug administration or apheresis within 20 days prior to the first IP administration.
14. Individuals who had received a blood transfusion within 30 days prior to study drug administration.
15. Exposure to any investigational drug within 6 months prior to the first IP administration.
16. Individuals taking any drugs inducing or inhibiting drug metabolizing enzymes including barbiturates within 30 days prior to the first IP administration.
17. Individuals who had consumed grapefruit juice > 5cups/day or caffeine > 5cups/day within 30 days prior to the first IP administration or who cannot stopping consume grapefruit juice or caffeine during clinical study.
18. Individuals who had drinking (alcohol > 30 g/day) within 30 days prior to the first IP administration or who cannot stopping drink.
19. Heavy smoking (more than 10 cigarettes/day) within 30 days prior to screening or who cannot quit smoking during clinical study.
20. Pregnant or women who may be pregnant
21. Subjects having been deemed inappropriate for the trial as determined by the investigator.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-501, D759, D150, CKD-393 | Time Frame: 0 hour ~ 48 hours
  Area under the CKD-501/D759/D150/CKD-393 concentration in blood-time curve from zero to final
Cmax of CKD-501, D759, D150, CKD-393 | Time Frame: 0 hour ~ 48 hours
  The maximum CKD-501/D759/D150/CKD-393 concentration in blood sampling time t

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No